CLINICAL TRIAL: NCT00660192
Title: Investigation of Efficacy and Safety of Botulinum Toxin A (Botox-Allergan Inc) in Migraine Headaches
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0709003056
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Refractory Migraine
Keywords: Migraine, refractory migraine, Pain, Botulinum Toxin , Botox
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects are randomized to receive Placebo which is inactive saline (sterile salt water solution). The Subjects are injected with a comparable amount of placebo solution (2cc-3cc) as received by those randomized to receive active study drug. The randomization will be done in a double blinded manner where the investigator nor the subject knows which substance (Placebo vs. Botox) is being injected.
  Interventions: Other: Placebo
- Botox (Active Comparator): Subjects are randomized to receive Active study drug Botox (onobotulinumtoxinA). The Botox is prepare by diluting 100units of toxin /1cc Saline. The Subjects are injected with 200-300units of units of Botox which is 2cc-3cc of solution. The randomization will be done in a double blinded manner where the investigator nor the subject knows which substance (Placebo vs. Botox) is being injected.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — subjects randomized to receive Botox with have a series of injections of onobotulinumtoxinA totalling 200 to 300 units. Botox is prepared b adding 1cc of preservative free saline in 100 unit vial. Final dose is determined by bod and neck size.
  Other Names: onobotulinumtoxinA
  Arms: Botox
Other: Placebo — subjects randomized to receive Placebo will have a series of injections of saline solution totalling 2cc's to 3cc's injected into the scalp in a halo pattern; and into affected neck muscles.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The hypothesis of this study is that injection of botulinum toxin A into the muscles around the head (frontal, temporal, posterior neck, occipital) can reduce the intensity and frequency of migraine headaches by 50%.

DETAILED DESCRIPTION:
Contact PI for study details

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* Migraine for more than three months, that fail to respond to two or more major anti-migraine drug, meeting criteria of chronic migraine

Exclusion Criteria:

* Age below 18
* Pregnant or may become pregnant
* Disease of neuromuscular junction or drugs that affect N-M junction
* Allergy to Botox
* Previous use of Botox for migraine by similar methodology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Jabbari, M.D., Principal Investigator — Yale- 203-737-2464
Locations (1):
- Yale Physician's Building, 800 Howard Ave, lower level,, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects randomized to placebo ho receive injections of 2cc's to 3cc's of saline solution. into muscle of the scalp and neck.
- Botox: Subjects randomized to receive 200-300units of onobotulinumtoxinA by injections into the scalp and neck muscles
Period: Overall Study
Arm/Group | Placebo | Botox
Started | 12 | 13
Completed | 10 | 10
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Botox | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Full Range); unit: years] | 59 [18 to 80] | 61 [18 to 80] | 60 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 7 | 13
Pain [Mean (Full Range); unit: units on a scale] — Pain score on the Visual Analog scale. VAS ranges from 0-10, with 0 being no pain, and 10 being worst pain.
  units on a scale | 8.1 [0 to 10] | 8.3 [0 to 10] | 8.24 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Days of Decrease in Pain Level Using VAS
Description: Number of days of decreased pain (2 grades or more) on Visual Analog scale. VAS ranges from 0-10, with 0 being no pain, and 10 being worst pain.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo: Inactive Saline
- Botullinum Toxin: Subjects injected with 100-200 units of botox depending on body and neck size
Arm/Group | Placebo | Botullinum Toxin
Number analyzed (Participants) | 10 | 10
days | 1.20 (5.63) | 8.67 (8.18)
Statistical Analysis 1: Comparison: Placebo vs Botullinum Toxin; Test type: Superiority or Other; p = 0.0347, t-test, 2 sided

2. Secondary Outcome: Number of Participants Satisfied With Treatment
Description: Number of Patients whose Patient global impression of change (PGIC) moderately or much improved- The PGIC is a 7 point scale that requires the clinician to assess how much the patient's pain has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:
  No change (or condition has gotten worse) (1) Almost the same, hardly any change at all (2) A little better, but no noticeable change (3) Somewhat better, but the change has not made any real difference (4) Moderately better, and a slight but noticeable change (5) Better and a definite improvement that has made a real and worthwhile difference (6) A great deal better and a considerable improvement that has made all the difference (7)improved
  This outcome is number of patients who chose a 6 or above on the PGIC 6 weeks after treatment.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Botullinum Toxin
Number analyzed (Participants) | 10 | 10
participants | 9 | 3
Statistical Analysis 1: Comparison: Placebo vs Botullinum Toxin; Test type: Superiority or Other; p = 0.0300, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Saline | Botox
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=12) | Botox (N=13)
Pain at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold symptoms (Infections and infestations) | 0 (0) | 1 (1) — Patient experienced colds symptoms 3-4 days after injection

LIMITATIONS AND CAVEATS:
Small study- results could have been different if numbers were larger Technique of injection different from PREEMPT study. Larger doses were injected into temporal and posterior neck muscles. No trapezius injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No